CLINICAL TRIAL: NCT06844435
Title: Continuous Renal Replacement Therapy (CRRT) in Surgery Room During Orthotopic Liver Transplantation (OLT)
Acronym: CRRT-OLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CRRT-OLT
Record Dates: First submitted 2024-12-03; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Liver Failure; Acute Kidney Injury; Kidney Disease, Chronic
Keywords: CRRT; Liver transplant
MeSH Terms: conditions — Liver Failure; Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: The study is aimed at analyzing the behavior of different indicators of clinical complications and comparing them with what was found in the historical series, in the hypothesis that with the new procedure the analyzed parameters are better.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CRRT during OLT (Other): CRRT during OLT
  Interventions: Other: continuous renal replacement therapy

INTERVENTIONS:
Other: continuous renal replacement therapy — continuous renal replacement therapy during OLT in surgery room

SUMMARY:
The study is interventional, non-pharmacological, single-center. The aim of this study is to test the possible added value of CRRT in the surgery room during liver transplantation, compared to the investigators center current practice in which CRRT is suspended and possibly restarted at the end of the operation. The incidence of some clinical and metabolic alterations that often complicate transplantation in the absence of CRRT will be evaluated, by measuring a series of parameters related to the state of water filling, acid-base balance, general metabolic structure, hemodynamics and supportive drugs.

Some parameters related to patient safety will be evaluated. The results of this exploratory study will be useful to document what was rationally hypothesized, that is, that the continuation of dialysis treatment even during the hours of surgery, in this narrow category of patients, is actually useful to reduce the possible clinical and metabolic complications, intra- and/or post-operative (within 48 hours of transplant), linked to the simultaneous presence of renal failure.

The statistical analysis is aimed at analyzing the behavior of different indicators of clinical complications and comparing them with what was found in the historical series, in the hypothesis that with the new procedure the analyzed parameters are better. In detail, the mean values at the end of treatment will be compared for:

* Central venous pressure
* Potassiemia
* Lactatemia
* pH

The following will also be evaluated:

* dose of vasoconstrictor drugs, defined by the variation between the dose at the beginning of administration during the anhepatic phase and the maximum dose reached
* pulmonary congestion/pulmonary edema, defined by radiological signs of alveolar congestion/edema on chest X-ray in the post-surgery period
* safety parameters: episodes of hypokalemia requiring supplementation (K<3.5 mmol/l), post-surgery hypophosphatemia, number of coagulation events in the extracorporeal circuit, appearance of cardiac arrhythmias.

DETAILED DESCRIPTION:
The study is interventional, non-pharmacological, single-center. The clinical practice adopted to date provides that upon arrival of the liver to be transplanted, dialysis is interrupted before entering the surgery room, and then resumed, if necessary, upon exiting the room. The aim of this study is to test the possible added value of CRRT in the surgery room during liver transplantation, compared to the investigators center current practice. The incidence of some clinical and metabolic alterations that often complicate transplantation in the absence of CRRT will be evaluated, by measuring a series of parameters related to the state of water filling, acid-base balance, general metabolic structure, hemodynamics and supportive drugs. Some parameters related to patient safety will be evaluated.

For each patient enrolled in the study, the following will be collected:

baseline data (taken before entering the operating room), intraoperative data, postoperative data for the first 48 hours, and data at 3 and 6 months after surgery.

Baseline data:

* demographic data: age, sex
* anamnestic data: etiology of liver disease (viral, alcoholic, neoplastic, other); state of liver disease (acute, acute on chronic, cirrhosis, decompensated cirrhosis); etiology of acute kidney injury (sepsis, hypovolemia/hemorrhage, iatrogenic/drugs, hepatorenal syndrome, other); indication for dialysis treatment (uremia, electrolyte imbalance, acidosis, oligo-anuria, fluid overload, other)
* biochemical parameters (as indicated in the "Objectives" paragraph): pH, HCO3, pO2, pCO2, BE, P/F ratio, DO2, SVO2; hemoglobin, hematocrit, sodium, potassium, calcium, lactate, CPK, ammonium, glycemia
* Hemodynamic parameters: heart rate, mean arterial pressure, cardiac output, peripheral vascular resistance, central venous pressure, pulmonary wedge pressure, stroke volume
* Severity scores: MELD and SOFA pre- and post-intervention
* Other clinical data: amine infusion (YES/NO), mechanical ventilation (YES/NO), urine output (volume/minute), radiological signs of pulmonary congestion/edema (YES/NO).

Intra- and post-operative data:

The biochemical, hemodynamic and clinical parameters listed above will be recorded at the following times:

* at the induction of anesthesia
* in the anhepatic phase
* at 5, 30 and 120 and 180 minutes after reperfusion
* at the end of surgery
* at 24 and 48 hours after leaving the operating room The following will also be reported: intraoperative onset of arrhythmia (YES/NO), intraoperative coagulation of the extracorporeal circuit (YES/NO), intraoperative replacement of the extracorporeal circuit for TMP>200 (YES/NO), onset of hypophosphatemia (<2.5 mg\dl) and hypocalcemia (calcium ion <0.9 mmol\l) hypercalcemia (calcium ion <1.3 mmol\l) assessed at the end of surgery.

Data 3 and 6 months post intervention:

* survival
* INR
* Bilirubin
* Creatinine
* GFR

CRRT protocol:

The extracorporeal renal function replacement treatment modality adopted in the population under study is continuous veno-venous hemodiafiltration (CVVHDF) without anticoagulation. The Prismax® Baxter monitor will be used. A commercially available dialysis solution will be used and in particular: Prismasol 2 ® Baxter used both as dialysate and as post-dilution reinfusion, blood flow 150 ml/min; dialysis dose initially prescribed 30-35 ml/min which may be increased during treatment if necessary to obtain better metabolic/electrolytic control.

During the transplant, a dialysis nurse will be present in the surgery room for the entire duration of the operation. At the end of the operation, CRRT will continue in Intensive Care Unit.

The results of this exploratory study will be useful to document what was rationally hypothesized, that is, that the continuation of dialysis treatment even during the hours of surgery, in this narrow category of patients, is actually useful to reduce the possible clinical and metabolic complications, intra- and/or post-operative (within 48 hours of transplant), linked to the simultaneous presence of renal failure.

The statistical analysis is aimed at analyzing the behavior of different indicators of clinical complications and comparing them with what was found in the historical series, in the hypothesis that with the new procedure the analyzed parameters are better. In detail, the mean values at the end of treatment will be compared for:

* Central venous pressure
* Potassiemia
* Lactatemia
* pH

The following will also be evaluated:

* dose of vasoconstrictor drugs, defined by the variation between the dose at the beginning of administration during the anhepatic phase and the maximum dose reached
* pulmonary congestion/pulmonary edema, defined by radiological signs of alveolar congestion/edema on chest X-ray in the post-surgery period
* safety parameters: episodes of hypokalemia requiring supplementation (K<3.5 mmol/l), post-surgery hypophosphatemia, number of coagulation events in the extracorporeal circuit, appearance of cardiac arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for ISOLATED LIVER TRANSPLANT with acute or chronic renal failure already undergoing continuous dialysis treatment in Intensive Care at the time of arrival of the organ. If acute renal failure: stage 2-3 of the KDIGO classification (referring to diuresis).
2. Patients scheduled for COMBINED LIVER-KIDNEY TRANSPLANT, whether or not they are already undergoing continuous dialysis treatment in Intensive Care at the time of arrival of the organ to be implanted
3. Patients scheduled for ISOLATED LIVER TRANSPLANT, for acute liver failure and with acute renal failure in stage 3 of the KDIGO classification (referring to diuresis) for which there is an indication for continuous dialysis.
4. Age ≥ 18 years
5. Signature of informed consent

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
central venous pressure average values at the end of treatment | during surgery
  Central venous pressure (cmH2O)
Potassiemia average values at the end of tretment | during surgery
  Potassiemia (mmol/L)
Lactatemia average values at the end of treatment | during surgery
  Lactatemia (mmol/L)
pH average values at the end of treatment | during surgery
  pH (absolute value)

SECONDARY OUTCOMES:
dose of vasocostrictors drugs | during surgery
  vasoconstrictor drugs, defined by the variation between the dose at the start of administration during the anhepatic phase and the maximum dose reached (mcg/Kg/min)
pulmunary congestion | during surgery
  pulmonary congestion/pulmonary edema, defined by radiological signs of alveolar congestion/edema on chest X-ray in the post-surgery period (Yes/NO)
safety parameters: episodes of hypokalemia | during surgery
  episodes of hypokalemia - K < 3.5 mmol/L - requiring supplementation (number of episodes)
safety parameters: post-surgery hypophosphatemia | during surgery
  onset of hypophosphatemia <2.5 mg\dl (Yes/No)
safety parameters: number of coagulation events in the extracorporeal circuit | during surgery
  intraoperative replacement of the extracorporeal circuit for TMP>200 (YES/NO)
Safety parameters: appearance of cardiac arrhythmias | during surgery
  appearance of cardiac arrhythmias (Yes/No)

OTHER OUTCOMES:
Survival at 3 and 6 months post intervention | 3 and 6 months post intervention
  Survival (Yes/No)
INR at 3 and 6 months post intervention | 3 and 6 months post intervention
  INR (International Normalized Ratio)
Bilirubin at 3 and 6 months post intervention | 3 and 6 months post intervention
  Bilirubin (mg/dL)
Serum Creatinine at 3 and 6 months post intervention | 3 and 6 months post intervention
  Serum Creatinine (mg/dL)
GFR at 3 and 6 months post intervention | 3 and 6 months post intervention
  GFR (mL/min/1.73 m2)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Ricci, Md, Phd, Principal Investigator — IRCCS Azienda ospedaliero-Universitaria di Bologna Policlinico di S'Orsola
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy